CLINICAL TRIAL: NCT05652127
Title: Examining the Impact of Child Mightier Play on Caregiver Stress and Wellbeing
Brief Title: Mightier Play and Caregiver Stress and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromotion Labs (Industry)
Responsible Party: Principal Investigator, Alyssa Peechatka, Lead Scientist, Neuromotion Labs
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NML-2109
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Stress
Keywords: Parent; Stress; Wellbeing

STUDY DESIGN:
Intervention Model Description: As a single arm study all participants' children will receive a game-based biofeedback intervention. They are encouraged to engage with the intervention in an entirely self-directed manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Child play of Mightier (Experimental): Ad lib child biofeedback video game play in home
  Interventions: Other: Mightier

INTERVENTIONS:
Other: Mightier — Mightier is an app-based biofeedback video game that utilizes heart rate (HR) monitoring during game play to teach and facilitate practice of emotional regulation skills in children ages 6-14

SUMMARY:
The primary goal of this study is to demonstrate that digital mental health interventions for children, such as Mightier, can have an impact on caregiver functioning, including parenting stress, overall wellbeing, and work engagement.

Participants will be caregivers of children who are using Mightier, a video-game based heart rate biofeedback intervention used to build emotion regulation. Caregivers will be asked to complete a short survey prior to their child's first play and then complete that survey two more times, at 8 weeks and 12 weeks post baseline.

The pre-post self report design will allow us to observe changes during Mightier use and relate those changes to overall engagement with the intervention.

DETAILED DESCRIPTION:
Providing care for children with mental illness is associated with significant caregiver burden that manifests in physical, psychological, and social ways. Caregiver burden is largely associated with child symptom severity. As such, reducing child symptom severity should reduce caregiver burden. Yet, caregiver burden is not commonly assessed as an outcome of mental health interventions and little is known about the impact of child-focused novel digital mental health interventions on caregiver burden.

Mightier is an app-based biofeedback video game platform that utilizes heart rate (HR) monitoring during game play to teach and facilitate practice of emotional regulation skills in children. The effectiveness of Mightier has been supported through several studies in children ages 8-18, specifically reducing symptoms of aggression, oppositional behavior, and parental stress. While prior work has supported that Mightier as a child-based intervention also decreases parent stress, we have not examined if child use of Mightier meaningfully impacts caregiver wellbeing, or if these changes translate to changes in work engagement or absenteeism. The proposed study will be a single arm trial where parents and caregivers who have purchased Mightier will complete baseline and follow up self-report measures assessing presenteeism, absenteeism, parenting stress, and overall wellbeing.

For this proposed study we hypothesize the following:

1. Participants will report significant reduction in parent stress and absenteeism and a significant increase in overall wellbeing and presenteeism.
2. Changes in participant stress will be negatively associated with child minutes of Mightier use and changes in participant wellbeing will be positively associated with child minutes of Mightier use.
3. Children of participants who report positive change in work productivity (increases in presenteeism or decreases in absenteeism) will have used Mightier significantly more than those who do not report positive change.

For the duration of the 8-12 week intervention period, participants will play Mightier and engage with Mightier parent content ad libitum. They will not receive any special instructions or recommendations outside of those provided to all Mightier families. Consistent with any other family using Mightier, participating families will be free to engage with or deny all programming associated with Mightier (e.g. email updates and other support). All individuals engaging with participating families to facilitate the standard Mightier experience will be blinded to their participation in research.

Participating families will be contacted via email to complete follow-up measures. These emails will be sent 1) 8 weeks after participants complete the first assessment and 2) 12 weeks after participants complete their first assessment. Participants will be sent the 12 week follow up email regardless of 8 week follow up assessment completion. Participants will only be sent these emails if they are customers of Mightier at the time of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregivers have a child engaging with the heart rate biofeedback intervention Mightier
* Parent or caregivers reside in the United States

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
Parental Stress Scale | 12 weeks
  The Parental Stress Scale is an 18-item questionnaire assessing parents' feelings about their parenting role, including both positive and negative aspects of parenthood. Scores range from 18 (lower stress) to 90 (higher stress).

SECONDARY OUTCOMES:
The Flourishing Scale | 12 weeks
  The Flourishing Scale is a brief 8-item measure of self-perceived success in important areas of functioning such as relationships, self-esteem, purpose, and optimism. Scores range from 8 to 56, where high scores represent greater levels of self-perceived success.
Caregiver work and valued activities engagement | 12 weeks
  1-5 items (depending on current employment status) measuring work absenteeism, work engagement, and valued activities engagement. The first question is an open ended numerical input of workdays missed to provide behavioral or mental health support to their child. The 4 following questions are Leikert-type questions ranging from strongly agree to strongly disagree, with strongly agree representing greater impairment of function. These questions have not been independently validated and are not a part of a formalized scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromotion Inc, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No